CLINICAL TRIAL: NCT01160809
Title: Effect of a Combined Use of Mosquito Repellent and Insecticide Treated Net on Malaria in Southern Ethiopia: a Cluster-randomized Controlled Trial
Brief Title: Effect of a Combined Use of Mosquito Repellent and Insecticide Treated Net on Malaria in Ethiopia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Malaria Consortium, Ethiopia (Other)
Collaborators: Addis Ababa University (Other); Columbia University (Other); Coalition Against Malaria in Ethiopia (Unknown)
Responsible Party: Dr. Wakgari Deressa, School of Public Health, Addis Ababa University, Ethiopia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0001
Record Dates: First submitted 2010-07-08; First posted 2010-07-12 (Estimated); Last update posted 2010-07-12 (Estimated); Status verified 2010-07

CONDITIONS: Malaria; Mosquito Repellent; Long Lasting Insecticidal Nets
Keywords: Malaria; Mosquito repellent; LLINs
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mosquito repellent and LLINs group vs. LLINs group only (Experimental): This study is based on two population groups: 1) a group of households that use LLINs alone (control) and 2) a group of households that use both mosquito repellent and LLINs (repellent group).
  Interventions: Other: Mosquito repellent

INTERVENTIONS:
Other: Mosquito repellent — Mosquito repellent (Buzz Off jelly) every evening applied to face, neck, hands and legs

SUMMARY:
The combined use of a mosquito repellent and long lasting insecticidal nets (LLINs) by household members would result in a 40% reduction in malaria prevalence compared with households that only use LLINs.

DETAILED DESCRIPTION:
It has been recognized that the use of malaria preventive measures in combination with LLINs could improve the effectiveness of nets in preventing the disease. This study examined the effect of a combined use of mosquito repellent (i.e., Buzz Off) and LLINs on malaria prevalence in an area of unstable and seasonal malaria transmission.

ELIGIBILITY:
Inclusion Criteria:

* All volunteer household members

Exclusion Criteria:

* Infants less than two months
* Not in the study area

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 6082 (Actual)
Dates: Start 2008-09; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Malaria parasite (P. falciparum and/or P. vivax)through microscopic detection
  The objective of the study is to investigate the impact of a combined use of mosquito repellent and LLINs in reducing malaria. The primary outcome of the study is detection of malaria parasites (P. falciparum and/or P. vivax) through examination of microscopic blood slides collected from finger-pricks.

SECONDARY OUTCOMES:
Household ownership and utilization of LLINs
  Owneship and utilization of LLINs by household members during the night before the baseline survey

CONTACTS AND LOCATIONS:
Locations (1):
- SNNPR, Ethiopia, Awasa, Snnpr, Ethiopia

REFERENCES:
- [Derived] Deressa W, Yihdego YY, Kebede Z, Batisso E, Tekalegne A, Dagne GA. Effect of combining mosquito repellent and insecticide treated net on malaria prevalence in Southern Ethiopia: a cluster-randomised trial. Parasit Vectors. 2014 Mar 28;7:132. doi: 10.1186/1756-3305-7-132. PMID 24678612